CLINICAL TRIAL: NCT02589106
Title: Safety and Efficacy of Anisotropic Textile Braces for Adolescent Idiopathic Scoliosis
Brief Title: Anisotropic Textile Braces for Adolescent Idiopathic Scoliosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Joanne Yip, Professor, The Hong Kong Polytechnic University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GRF2016
Record Dates: First submitted 2015-10-27; First posted 2015-10-28 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Scoliosis
Keywords: Anisotropic Textile Braces
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Anisotropic Textile Braces (Experimental): The design of the anisotropic textile braces will provide different mechanisms with rigid, semi-rigid and flexible materials: a) axial elongation through a close fit of the brace supported with textile composites on the lateral sides of the trunk, b) 3-point pressure with push and counter-pushes through semi-rigid pads inserted inside the pocket lining, c) pulling or compression to correct kyphosis or lordosis in the sagittal plane with elastic bands, d) derotation between the pelvis and shoulders with uneven straps, and e) an active mechanism with sensors added to the brace to maintain correct posture.
  Interventions: Device: Anisotropic Textile Braces

INTERVENTIONS:
Device: Anisotropic Textile Braces — The period of the wear trial is 12-18 months in time for each subject. Wear instructions (23 hrs per day) and wash instructions will be provided to the subjects before the wear trial. Evaluation tests based on health in consideration of the use of the anisotropic textile brace (heart and pulmonary function testing and sensory level measurements) will be carried out at the beginning of the wear trial. Clinical, radiography, self-report and follow-up after completion of the study

SUMMARY:
One of the most common types of 3-dimensional spinal deformities with unknown etiology in youths is adolescent idiopathic scoliosis (AIS). The spinal curvature increases as puberty progresses. Generally, rigid orthotic bracewear is prescribed as non-invasive treatment for moderate AIS if treatment begins early and the orthosis is worn with compliance. Obviously, teenage patients are reluctant to accept a rigid orthosis due to aesthetics and the physical constraint. Therefore, semi-rigid and flexible orthoses have been developed, but their efficacy is still controversial and there are other issues, such as high pain scores. There is clearly room for improvement. Therefore, a garment-type of bracewear will be designed and developed to correct spinal deformity, reduce the possibility of spinal curve progression, and satisfy the needs of the patients as well as take their psychological concerns into consideration.

DETAILED DESCRIPTION:
The design of the anisotropic textile braces will provide different mechanisms with rigid, semi-rigid and flexible materials:

1. axial elongation through a close fit of the brace supported with textile composites on the lateral sides of the trunk,
2. 3-point pressure with push and counter-pushes through semi-rigid pads inserted inside the pocket lining,
3. pulling or compression to correct kyphosis or lordosis in the sagittal plane with elastic bands,
4. derotation between the pelvis and shoulders with uneven straps, and
5. an active mechanism with sensors added to the brace to maintain correct posture.

ELIGIBILITY:
Inclusion Criteria:

* Aged 10 to 14 years
* Diagnosis of AIS
* a Cobb's angle between 20 to 30 degrees
* a Risser grade of the iliac crest of ≤ 2
* Pre-menarche or post- menarche by no more than 1 year
* Ability to read and understand English or Chinese
* Physical and mental ability to adhere to anisotropic textile braces protocol

Exclusion Criteria:

* Contraindications for x-ray exposure
* Diagnosis of other musculoskeletal or developmental illness that might be responsible for the spinal curvature
* History of previous surgical or orthotic treatment for AIS
* Contraindications for pulmonary and/ or exercise tests
* Psychiatric disorders
* Recent trauma
* Recent traumatic (emotional) event

Ages: 10 Years to 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression of the spinal curve | 18 months
  The spinal curve is said to be under control if the increase in the Cobb's angle is <5°

SECONDARY OUTCOMES:
Posture improvement | 18 months
  Improvement of posture by clinical photographs assessment

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The Hong Kong Polytechnic University, Hong Kong, Guangdong
  - The Hong Kong Polytechnic University, Hong Kong